CLINICAL TRIAL: NCT00986661
Title: A Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics of PV-10 Chemoablation of Cancer Metastatic to the Liver or Hepatocellular Carcinoma Not Amenable to Resection or Transplant
Brief Title: A Study to Assess PV-10 Chemoablation of Cancer of the Liver
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Provectus Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Provectus Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV-10-LC-01
Record Dates: First submitted 2009-09-24; First posted 2009-09-30 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Cancer Metastatic to the Liver; Hepatocellular Carcinoma; Metastatic Melanoma; Metastatic Ocular Melanoma; Metastatic Uveal Melanoma; Metastatic Lung Cancer; Metastatic Colon Cancer; Metastatic Colorectal Cancer; Metastatic Breast Cancer; Metastatic Pancreatic Cancer
Keywords: melanoma; uveal; ocular; mUM; mOM; OM; UM; pancreatic; colon; colorectal; lung; metastatic; carcinoid; neuroendocrine; liver; hepatic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Melanoma; Uveal Melanoma; Lung Neoplasms; Colonic Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Carcinoid Tumor | interventions — Rose Bengal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PV-10 Injection (Intralesional) (Experimental): Subjects in each of three cohorts will receive a single dose of PV-10 to one Target Lesion.
  Interventions: Drug: PV-10 (10% rose bengal disodium)

INTERVENTIONS:
Drug: PV-10 (10% rose bengal disodium) — Subjects will receive a single injection of PV-10 to a single Target Lesion (0.25 mL PV-10 per cc lesion volume, Lv, or 0.50 mL PV-10 per cc Lv).

SUMMARY:
This open-label study will evaluate the safety, tolerability, pharmacokinetics and effect on tumor growth following a single intralesional injection of PV-10 in subjects with either (a) hepatocellular carcinoma (HCC) that is not amenable to resection, transplant or other potentially curative therapy or (b) cancer metastatic to the liver.

DETAILED DESCRIPTION:
Subject will be enrolled in one of four planned cohorts (Main Study Group, Expansion Cohort 1, Expansion Cohort 2 or Expansion Cohort 3).

Main Study Group. Three initial subjects with either HCC or cancer metastatic to the liver will receive 0.25 mL PV-10 per cc lesion volume (Lv) to a single lesion (up to a maximum dose of 7.5 mL PV-10). If none of the initial three subjects experiences a new and persistent CTCAE Grade 3 or greater non-hematological or any Grade 4 hematological toxicity over a 28-day follow-up interval, an additional three subjects will be enrolled and similarly treated with PV-10 administered at 0.50 mL per cc Lv (up to a maximum dose of 15 mL PV-10) provided no new and persistent Grade 3 or greater non-hematological or any Grade 4 hematological toxicity occurs.

Expansion Cohort 1 (EC1: PV-10 plus/minus Checkpoint Inhibition). Following demonstration of safety and tolerability in the Main Study Group, up to 48 additional subjects with cancers metastatic to the liver or with HCC will be enrolled into Expansion Cohort 1 (EC1). Subjects will be treated with PV-10 administered at 0.50 mL per cc Lv (up to a maximum dose of 15 mL PV-10). Subjects may receive injection of up to two lesions in any PV-10 treatment cycle. Enrollment will continue provided no new and persistent Grade 3 or greater non-hematological (excluding fatigue) or any Grade 4 hematological toxicity occurs.

Expansion Cohort 2 (EC2: PV-10 plus Checkpoint Inhibition). Following demonstration of safety and tolerability in the Main Study Group, up to 12 additional subjects with HCC on a background of standard care checkpoint inhibition therapy (i.e., anti-PD-1 therapy) will be enrolled into Expansion Cohort 2 (EC2). Subjects will be treated with PV-10 administered at 0.50 mL per cc Lv (up to a maximum dose of 15 mL PV-10). Subjects may receive injection of up to two lesions in any PV-10 treatment cycle. Enrollment will continue provided no new and persistent Grade 3 or greater non-hematological (excluding fatigue) or any Grade 4 hematological toxicity occurs.

Expansion Cohort 3 (EC3: PV-10 plus Checkpoint Inhibition). Following demonstration of safety and tolerability in the Main Study Group, up to 12 additional subjects with hepatic metastases of uveal melanoma (mUM) on a background of standard care checkpoint inhibition therapy (i.e., anti-CTLA-4, anti-PD-1 or combination anti-CTLA-4 and anti-PD-1 therapy) will be enrolled into Expansion Cohort 3 (EC3). Subjects will be treated with PV-10 administered at 0.50 mL per cc Lv (up to a maximum dose of 15 mL PV-10). Subjects may receive injection of up to two lesions in any PV-10 treatment cycle. Enrollment will continue provided no new and persistent Grade 3 or greater non-hematological (excluding fatigue) or any Grade 4 hematological toxicity occurs.

Concomitant therapy with immune checkpoint inhibition is allowed in Expansion Cohort 1 and required in Expansion Cohort 2 and Expansion Cohort 3. This concomitant therapy must commence at least 7 days prior to initial PV-10 administration.

Subjects in each Expansion Cohort one or more additional injectable tumor ≥ 1 cm in diameter will be eligible for treatment of one or more additional injectable tumor 28 days to 6 months after prior PV-10 administration provided that any prior treatments with PV-10 were well tolerated. This may be repeated until all injectable tumors ≥ 1 cm in diameter have received PV-10.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, males and females.
* Histologically or cytologically confirmed, or clinically diagnosed based on currently accepted standards, cancer metastatic to the liver or HCC that is not amenable at the time of enrollment to resection, transplant or other potentially curative therapy.
* At least one Target Lesion determined to be amenable to percutaneous injection by the treating physician.
* Target Lesion(s) must have measurable disease, defined as a unidimensionally measurable lesion ≥ 1.0 cm in longest diameter by helical CT; the maximum diameter of Target Lesion(s) shall be ≤ 4.9 cm.
* Performance status of Karnofsky scale 60%-100% or ECOG performance scale 0-2.
* Life expectancy ≥ 12 weeks.
* Hematopoietic Function: WBC ≥ 2,500/mm3; ANC ≥ 1000/mm3; Hemoglobin ≥ 8 g/dL; Platelet count ≥ 50,000/mm3; Coagulation: INR ≤ 1.3.
* AST and ALT < 5 times ULN; ALP < 5 times ULN; Bilirubin ≤ 1.5 times ULN; Creatinine ≤ 1.5 times ULN and eGFR ≥ 50.
* Thyroid Function: Total T3 or free T3, total T4 or free T4 and THS ≤ CTCAE Grade 2 abnormality.
* Renal Function: Adequate renal function in the opinion of the Investigator with no clinically significant renal impairment or uncontrolled renal disease.
* Cardiovascular Function: Adequate cardiovascular function in the opinion of the Investigator with no clinically significant uncontrolled cardiovascular disease.
* Respiratory Function: Adequate respiratory function in the opinion of the Investigator with no clinically significant uncontrolled respiratory disease.
* Immunological Function: Adequate immune system function in the opinion of the Investigator with no known immunodeficiency disease.
* Informed Consent: Signed by the subject prior to screening.

Exclusion Criteria:

* Target Lesion(s) must not be contiguous with, encompass or infiltrate major blood vessels.
* Primary HCC amenable to resection, transplant or other potentially curative therapy.
* Surgery: Subjects who have received hepatic surgery, ablation or chemoembolization within 4 weeks of PV-10 administration.
* Radiation Therapy: Hepatic radiation within 4 weeks of PV-10 administration.
* Chemotherapy: Chemotherapy within 4 weeks of PV-10 administration (6 weeks for nitrosoureas or mitomycin C).
* Investigational Agents: Investigational agents within 4 weeks (or 5 half-lives) of PV-10 administration.
* Phototoxic or Photosensitizing Agents: Concomitant agents posing a clinically significant risk of photosensitivity reaction within 5 half-lives of PV-10 administration.
* Concurrent or Intercurrent Illness: Impaired wound healing due to diabetes; Significant concurrent or intercurrent illness, psychiatric disorders or alcohol or chemical dependence that would compromise Subject safety or compliance or interfere with interpretation of the study; Uncontrolled thyroid disease or cystic fibrosis; Presence of clinically significant acute or unstable cardiovascular, cerebrovascular (stroke), renal, gastrointestinal, pulmonary, immunological (with the exception of the presence of hepatitis B virus (HBV), viral hepatitis, or cirrhosis), endocrine, or central nervous system disorders; Current encephalopathy or current treatment for encephalopathy; Variceal bleeding requiring hospitalization or transfusion within 4 months of screening; History of human immunodeficiency virus or acquired immune deficiency syndrome; The clinical presence of ascites.
* Pregnancy: Female subjects who are pregnant, lactating or have positive serum β HCG pregnancy test taken within 7 days of PV-10 administration; Fertile subjects who are not using effective contraception (e.g., oral contraceptives, intrauterine devices, double barrier methods such as condoms and diaphragms, abstinence or equivalent measures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2009-10; Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of hepatic administration of PV-10 | 28 days
  Systemic and locoregional Adverse Events (AEs) will be graded by CTCAE v4.0 and coded according to MedDRA; AE data for all subjects in the 1st cohort will be assessed prior to dose escalation. Final assessment use AE data for all subjects

SECONDARY OUTCOMES:
PV-10 distribution | 3 months
  Lesion distribution and retention of PV-10 following injection assessed by CT
Objective response rate (ORR) | 3 months
  Objective response rate (ORR) of Target and measurable Bystander Lesions (if present) by 2D EASL and/or RECIST criteria
Changes in markers of hepatic function | 3 months
  Changes in markers of hepatic function, including ALP, ALT, AST, total bilirubin
Pharmacokinetics of PV-10 | 28 days
  Pharmacokinetics of PV-10 in the bloodstream following intralesional injection; samples will be obtained immediately prior to PV-10 injection and at 2, 4, 8, 24 and 72 hours, and 7, 14 and 28 days to assess uptake and excretion of PV-10
Overall survival | Assessed every 3 months for up to 100 months
  Overall survival will be assessed for the intent-to-treat population

OTHER OUTCOMES:
Exploratory Correlative Endpoints | 28 days
  Serial correlative samples may be collected from subjects in each Expansion Cohort to evaluate potential changes in subjects' immunologic activity in response to PV-10 treatment; samples will be analyzed at one or more Sponsor-designated central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, PhD, Study Director — Provectus Biopharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Sharp Memorial Hospital, San Diego, California
  - Florida Hospital Tampa, Tampa, Florida
  - St Luke's University Health Network, Bethlehem, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas